CLINICAL TRIAL: NCT04969835
Title: A Phase 1, Open Label, Dose-Escalation and Expansion Study to Evaluate the Safety, Pharmacokinetics and Initial Therapeutic Activity of AVA6000, a Novel FAP-activated Doxorubicin Administered Intravenously in Patients With Locally Advanced or Metastatic Selected Solid Tumours
Brief Title: A Study Evaluating the Safety, Pharmacokinetics and Early Efficacy of AVA6000 in Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Avacta Life Sciences Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALS-6000-101
Record Dates: First submitted 2021-06-22; First posted 2021-07-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Salivary Gland Tumor; Urothelial Carcinoma; Ovarian Carcinoma; Breast Cancer; Soft Tissue Sarcoma
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Transitional Cell; Ovarian Neoplasms; Breast Neoplasms; Sarcoma

STUDY DESIGN:
Intervention Model Description: This study will follow a standard 3+3 dose escalation design in Phase 1a to evaluate the safety, tolerability, and MTD of two AVA6000 administration schedules (Q3W and Q2W). The Phase 1b dose expansion regimen was selected based upon completion of the Phase 1a portion. A cohort at RDE -1 was added to select the optimal biologic dose. Cardiac safety will be assessed at cumulative exposure above the standard lifetime maximum exposure of doxorubicin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AVA6000 Phase 1a Dose Escalation Q3W (Experimental): Patients in this arm will receive escalating doses of AVA6000 following a 3+3 design, Q3W until disease progression, unacceptable toxicities, withdrawal from treatment for other reasons, reaching maximum lifetime cumulative exposure to doxorubicin (or other anthracyclines), or death, whichever occurs first.
  Interventions: Drug: AVA6000
- AVA6000 Phase 1a Dose Escalation Q2W (Experimental): Patients in this arm will receive escalating doses of AVA6000 following a 3+3 design, Q2W until disease progression, unacceptable toxicities, withdrawal from treatment for other reasons, reaching maximum lifetime cumulative exposure to doxorubicin (or other anthracyclines), or death, whichever occurs first.
  Interventions: Drug: AVA6000
- AVA6000 Phase 1b Dose Expansion (Experimental): Patients in this arm will receive AVA6000 at the recommended dose for expansion, until disease progression, unacceptable toxicities, withdrawal from treatment for other reasons, or death, whichever occurs first.
  Interventions: Drug: AVA6000
- AVA6000 Phase 1b Dose Expansion (dose identification) (Experimental): Dosing on this arm will occur at RDE -1 to identify the optimal biologic dose of AVA6000. Patients on this arm will receive AVA6000 until disease progression, unacceptable toxicities, withdrawal from treatment for other reasons, or death, whichever occurs first.
  Interventions: Drug: AVA6000

INTERVENTIONS:
Drug: AVA6000 — AVA6000 is a FAP-activated doxorubicin.

SUMMARY:
This is a first-in-human (FIH), Phase 1 open-label, multicentre dose escalation study investigating AVA6000 monotherapy administered intravenously in patients with locally advanced (unresectable) or metastatic solid tumours that are likely to be FAP positive. The study consists of an initial Phase 1a dose escalation portion and a subsequent Phase 1b dose expansion portion upon completion of the dose escalation portion.

DETAILED DESCRIPTION:
Phase 1a (Dose Escalation): The dose-escalation portion is designed to evaluate the safety, tolerability and MTD and/or RP2D of AVA6000, administered as monotherapy in two schedules: Day 1 of a 21-day cycle (Q3W schedule) and Day 1 of a 14-day cycle (Q2W schedule).

Phase 1b (Dose Expansion): The dose-expansion arm is based on review of data in the dose escalation phase, with AVA6000 administered at the recommended dose for expansion.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has been fully informed about the study and has signed the Informed Consent Form.
2. Male or female patients, ≥ 18 years of age.
3. a) Phase 1a: patients with tumours reported to be FAP positive with histological or cytological confirmation of a locally advanced (unresectable) and/or metastatic:

   a. salivary gland, urothelial, ovarian, or breast carcinoma, who have either relapsed or progressed on SoC treatment or are intolerant or nonamenable to SoC treatment; OR b. soft-tissue sarcoma who: i. is treatment naïve in the locally advanced (unresectable) or metastatic setting and anthracycline naïve (any setting) and would otherwise be a candidate for doxorubicin hydrochloride treatment; OR ii. has received a total doxorubicin dose of < 150mg/m2 (any setting (< 2 cycles of 75 mg/m2 Q21 days) and has discontinued due to intolerance or toxicity related to doxorubicin

   b) Phase 1b: patients with histological or cytological confirmation of a locally advanced (unresectable) and/or metastatic tumour of one of the following types:
   1. High grade soft tissue sarcoma: histologically proven locally advanced or metastatic, unresectable progressive or recurrent DDLS or UPS who have received 0 or 1 prior lines of therapy in the locally advanced or metastatic setting
   2. SGC: Locally advanced or metastatic salivary gland confirmed by histopathology that cannot be completely resected by surgery who have received 0 or 2 prior lines of therapy in the locally advanced or metastatic setting. In addition, patients with adenoid cystic carcinoma subtypes must not have received prior cytotoxic therapy for locally advanced or metastatic disease. Adenoid cystic carcinoma subtype may be capped at 15 patients (assuming cohort of approximately 30 patients)
   3. TNBC: Locally advanced or metastatic triple negative breast cancer confirmed by histopathology who have received any prior therapy in the locally advanced or metastatic setting. Patients must be BRCA wild-type.
4. In Phase 1b, patients must meet the following additional criteria:

   Patients must demonstrate (as documented, per the investigator's assessment), radiological disease progression over the 6 months (±2 months) prior to screening. However, this requirement does not apply if the patient is newly diagnosed, recurrent or newly metastatic.
   * Patients must have measurable disease per RECIST.
   * Patients with high grade soft tissue sarcoma or salivary gland cancer must not have previously received an anthracycline-based therapy.
   * Patients with TNBC may receive up to 250mg/m2 of prior doxorubicin (or an equivalent anthracycline). Prior anthracycline based therapy must have been completed at least 6 months before the planned Cycle 1 Day 1 AVA6000 infusion. Prior anthracycline use must have been in the adjuvant or neoadjuvant setting only.
   * Patients must provide at least 1 tissue sample collection, either archival or fresh tissue (approximately 10 slides) unless the biopsy is medically not able to be performed or the principal investigator deems it is not medically feasible.
5. Has a life expectancy of ≥12 weeks, in the opinion of the investigator.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
7. Has recovered from all acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure (must have resolved to CTCAE grade ≤1 or returned to baseline, except alopecia and peripheral neuropathy, which can be up to CTCAE grade 2).
8. Has adequate haematological function (applies only to patients not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose):

   * Absolute Neutrophil count (ANC) of ≥1.5 × 109 cells/L.
   * Haemoglobin ≥9.0 g/dL.
   * Platelet count of ≥75,000/µL.
   * International normalised ratio (INR) and activated partial thromboplastin time (aPTT) ≤1.5 times the upper limit of normal (ULN).
9. Has adequate liver function:

   * Total bilirubin below ULN (except for patients with Gilbert's Syndrome who must have a total bilirubin <3 × ULN).
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (in patients with liver metastases, <5 × ULN is allowed).
   * Alkaline phosphatase (ALP) <5 × ULN in patients with documented liver or bone metastases, or ALP < 2 × ULN in patients without documented metastases.
10. Has adequate renal function (creatinine clearance ≥50 mL/min by Cockcroft-Gault formula) or patients with normal plasmatic creatinine despite creatinine clearance < 50 mL/min as per Cockcroft-Gault formula are eligible for the study.
11. Women of childbearing potential (WOCBP) and women who have ≤ 2 years amenorrhea after start of menopause: has a negative serum pregnancy test within 7 days prior to Cycle 1 Day 1.
12. Contraception requirements:

    * Female patients of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method (Pearl Index failure rate <1% per year) during the treatment period and for at least 6 months after the last dose of study drug.
    * Male patients with female partners of childbearing potential must agree to using 2 acceptable methods of contraception (Pearl Index failure rate <1% per year), including a barrier method (with or without spermicide) during the treatment period and for at least 6 months after the last dose of study drug.
    * Male patients must agree to refrain from sperm donation during the treatment period and for at least 6 months after the last dose of study drug.
13. All patients should have peripheral veins or central line that are, in the opinion of the Investigator or delegate, suitable for peripheral or central intravenous infusion of AVA6000.
14. The patient is willing and able to comply with the protocol, including any PK blood sampling requirements and agrees to return to hospital for follow-up visits and examinations.

Exclusion Criteria:

1. Has received trastuzumab within 7 months of the planned Cycle 1 Day 1 AVA6000 infusion.
2. Has received a prior total cumulative anthracycline dose of ≥ 350 mg/m2 doxorubicin (or equivalent anthracycline dose).
3. Has clinically significant or untreated central nervous system (CNS) metastases or leptomeningeal disease requiring treatment, as determined by the Investigator.
4. Patients who have any history of an active (requiring treatment) other malignancy (except any in-situ carcinoma, non-melanoma skin carcinoma and early prostate cancer with a normal PSA) within 2 years of study entry.
5. Has a significant, uncontrolled, concomitant disease that could affect compliance with the protocol.
6. In the opinion of the investigator, has uncontrolled hypertension (systolic blood pressure >150 mm Hg and/or diastolic blood pressure >100 mm Hg), unstable angina, CHF (New York Heart Association (NYHA) Class >II), left ventricular ejection fraction (LVEF) <55% or the low limit of institutional normal limit (whichever is lower) by echocardiogram (ECHO), serious cardiac arrhythmia requiring treatment (exceptions include atrial fibrillation, paroxysmal supraventricular tachycardia), history of myocardial infarction within 6 months prior to Cycle 1 Day 1, or history of uncontrolled cardiovascular disease or high-sensitivity troponin above normal at baseline (T or I).
7. Has a screening baseline mean corrected QTcF interval by Fridericia (QTcF) of >480 msec. Electrocardiograms (ECGs) will be evaluated locally at the investigator site. Has any clinically significant abnormalities in rhythm, conduction, or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec). Has any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, known family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval, a baseline resting bradycardia <45 beats/min or a baseline resting tachycardia of >100 beats/min.
8. HIV infection:

   * Patients with an AIDS-defining infection within 12 months of planned study Day 1.
   * Patients on anti-retroviral treatment who are not established on anti-retroviral treatment for ≥4 weeks and who have a viral load > 400 copies/mL prior to study Day 1.
9. Active hepatitis B (HBV) or hepatitis C (HCV) infection defined as:

   1. Has a positive hepatitis B surface antigen (HBsAG) test at screening. Patients with a past or resolved HBV infection (defined as having a negative HBsAG test and a positive antibody to hepatitis B core antigen [antiHBc] antibody test) are eligible.
   2. Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
   3. Chronic HBV (HbSAg positive, undetectable or low HBV DNA and normal ALT).
   4. Patients with active disease who have not on/initiated anti-retroviral treatment prior to study Day 1.
   5. Patients with untreated HCV infection or have not completed treatment for HCV infection.
   6. Patients with treated HCV infection but with a HCV viral load above the level of quantification.
10. Has a severe infection (requiring iv treatment) within 21 days prior to Cycle 1, Day 1 including, but not limited to, hospitalisation for complications of infection, bacteraemia, or severe pneumonia.
11. Has any other clinically significant active disease, metabolic dysfunction, physical examination finding, clinical laboratory finding, or reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Up to 28 days after the first dose of study therapy
  Incidence and nature of DLTs
Adverse events (AEs) | From Day 1 until up to 30 days after last dose of study drug.
  Incidence and severity of treatment-emergent (TE) and treatment-related adverse events (TRAEs) and Seious Adverse Events (SAEs).
Laboratory abnormalities | From Day 1 until up to 30 days after last dose of study drug.
  Incidence of clinically significant laboratory abnormalities and changes in laboratory values (haematology, coagulation, serum chemistry and urinalysis).
Vital signs | From Day 1 until up to 30 days after last dose of study drug.
  Clinically significant changes in vital signs, physical examination findings, and ECG findings.
Cardiac safety | From Day 1 until up to 30 days after last dose of study drug.
  Clinically significant reduction in LVEF (fallen by > 10% to below the lower level of institutional normal (as assessed by ECHO).

SECONDARY OUTCOMES:
Maximum drug concentration (Cmax) of AVA6000 & Doxorubicin | Cycle 1 and Cycle 2, 0-72 hours post dose (Dose Escalation)
  Cmax (maximum plasma concentration) of AVA6000 and Doxorubicin after administration after Cycle 1 and 2 for 72 hours post-dose.
Area under the curve (AUC) of AVA6000 & Doxorubicin | Cycle 1 and Cycle 2, 0-72 hours post dose (Dose Escalation)
  AUC (Area under the curve) of AVA6000 and Doxorubicin after administration after Cycle 1 and 2 for 72 hours post-dose.
Elimination half-life (t1/2) of AVA6000 & Doxorubicin | Cycle 1 and Cycle 2, 0-72 hours post dose (Dose Escalation)
  t1/2 (Elimination half-life) of AVA6000 and Doxorubicin after administration after Cycle 1 and 2 for 72 hours post-dose.
Renal clearance (CLr) of AVA6000 & Doxorubicin | Cycle 1 and Cycle 2, 0-72 hours post dose (Dose Escalation)
  CLr (Renal clearance) of AVA6000 and Doxorubicin after administration after Cycle 1 and 2 for 72 hours post-dose.
Objective response rate (ORR) | Up to one year
  ORR is defined as the proportion of patients achieving a best overall response of confirmed partial responses (PR) or complete response (CR), per Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
Duration of Response (DoR) | Up to one year
  DoR is defined as the duration of time from date of first response to date of disease progression, as per RECIST v1.1
Progression-free-survival (PFS) | Up to one year
  PFS is defined as the time from the date of the first dose to the date of the first documentation of confirmed disease progression or death, whichever occurs first, as per RECIST v1.1
Overall survival (OS) | Up to one year
  Overall survival (OS), defined as the date of first dose) to the occurrence of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Chris Twelves, MD, Principal Investigator — St James's University Hospital, Leeds, UK
Locations (9):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- United Kingdom (6):
  - The Beatson West of Scotland Cancer Centre, NHS Greater Glasgow & Clyde, Glasgow
  - St James's University Hospital, The Leeds Teaching Hospitals NHS Trust, Leeds
  - The Royal Marsden, NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Freeman Hospital, Newcastle-upon-Tyne NHS Foundation Trust, Newcastle upon Tyne
  - Weston Park Cancer Centre, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient-level data through clincialtrials@avacta.com